CLINICAL TRIAL: NCT02665273
Title: A Randomized, Sham-controlled Trial of Greater Occipital Nerve Block as Second Line Therapy for ED Patients With Acute Migraine
Brief Title: Greater Occipital Nerve Block With Bupivacaine for Acute Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, PI, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-4754
Record Dates: First submitted 2016-01-15; First posted 2016-01-27 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Greater occipital nerve block (Experimental): Bilateral greater occipital nerve block with 3cc of 0.5% bupivacaine, delivered using fan technique
  Interventions: Procedure: Greater occipital nerve block
- Sham (Sham Comparator): Bilateral intradermal injection of 0.5cc of 0.5% bupivacaine, delivered superficially to the area overlying the greater occipital nerve
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Procedure: Greater occipital nerve block — Bilateral greater occipital nerve block
  Arms: Greater occipital nerve block
Drug: Bupivacaine — 0.5 cc of 0.5% bupivacaine injected intradermally
  Arms: Sham

SUMMARY:
This is a randomized, sham-controlled study of greater occipital nerve block (GONB) using bupivacaine 0.5% for emergency department patients with acute migraine. Patients are only enrolled if they fail first line therapy with metoclopramide.

DETAILED DESCRIPTION:
The investigators are testing the following hypothesis:

In a population of patients who present to an ED with acute migraine and have been treated with parenteral metoclopramide unsuccessfully, bilateral greater occipital nerve blocks with bupivicaine will provide greater rates of short-term and sustained headache freedom than bupivacaine injected intradermally.

ELIGIBILITY:
Inclusion Criteria:

* ED patient with acute migraine or probable migraine
* Fail first line therapy with metoclopramide

Exclusion Criteria:

* Can't obtain consent
* Concern for secondary headache
* Skull defect
* Propensity for bleeding
* Overlying infection
* Pregnancy
* Allergy, intolerance study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Greater Occipital Nerve Block | Sham
Started | 13 | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Greater Occipital Nerve Block | Sham | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10) | 40 (12) | 38 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 1 | 3 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28
Duration of headache [Median (Inter-Quartile Range); unit: hours] | 96 [60 to 160] | 48 [24 to 100] | 72 [24 to 120]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieve Freedom From Headache
Description: Pain assessed using a standard ordinal headache intensity scale, in which subjects describe their headache as "severe", "moderate", "mild", or "none". Those with headache level = none, experience freedom from headache.
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Greater Occipital Nerve Block | Sham
Number analyzed (Participants) | 13 | 15
Participants | 4 | 0

2. Secondary Outcome: Sustained Headache Relief
Description: Attaining a headache level of "mild" or "none" within one hour of procedure and maintaining this for 48 hours without use of additional medication
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Greater Occipital Nerve Block | Sham
Number analyzed (Participants) | 13 | 15
Participants | 3 | 0

3. Secondary Outcome: Would Want the Same Treatment Again During a Subsequent Migraine
Description: Participants will be asked the following question: Do you want to receive the same procedure the next time you come to the ER with migraine?
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Greater Occipital Nerve Block | Sham
Number analyzed (Participants) | 13 | 15
Participants | 5 | 3

4. Other Pre Specified Outcome: Change in Pain Score Assessed by Verbal Pain Scale (0-10)
Description: The numerical scale, 0-10 pain scores will be obtained with 0 being "no pain" and 10 being "the worst pain imaginable."
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Greater Occipital Nerve Block | Sham
Number analyzed (Participants) | 13 | 15
units on a scale | 3.3 (2.8) | 5.5 (2.4)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Greater Occipital Nerve Block | Sham
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 3/13 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Greater Occipital Nerve Block (N=13) | Sham (N=15)
injection site reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT02665273/Prot_SAP_000.pdf